CLINICAL TRIAL: NCT04087707
Title: A Clinical Pharmacological Study of TS-142 in Non-Elderly and Elderly Healthy Participants (A Repeated-Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of TS-142 in Elderly and Non-Elderly Participants)
Brief Title: Safety, Pharmacokinetic, and Pharmacodynamic Study of TS-142 in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS142-202
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Step1; No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Step 1;TS-142 (Experimental)
  Interventions: Drug: Step 1: TS-142
- Step 2;TS-142 (Experimental)
  Interventions: Drug: Step 2: TS-142; Drug: Step 2: Placebo
- Step 2;Placebo (Placebo Comparator)
  Interventions: Drug: Step 2: TS-142; Drug: Step 2: Placebo

INTERVENTIONS:
Drug: Step 1: TS-142 — Non-elderly participants will receive 20 mg of TS-142 once daily for 7 consective days
  Arms: Step 1;TS-142
Drug: Step 2: TS-142 — Elderly participants will receive 20 mg of TS-142 once daily for 7 consective days
  Arms: Step 2;Placebo; Step 2;TS-142
Drug: Step 2: Placebo — Elderly participants will receive placebo once daily for 7 consective days
  Arms: Step 2;Placebo; Step 2;TS-142

SUMMARY:
The purpose of this study is to investigate the safety, pharmacokinetics, and pharmacodynamics of repeated dosing of TS-142 when administered once daily to healthy Japanese non-elderly and elderly participants

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 and <25.0 kg/m^2 and body weight is more than 40.0 kg at screening inspection
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of clinically relevant disease of any organ system that may interfere with the objectives of the study or provide a risk to the health of the participant
* History of drug and food allergy
* Other protocol defined exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) | Day 1 up to Day 14
  Number of Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) reported as mild, moderate, severe
Area under the concentration-time curve AUC (tau) | Day 1 up to Day 9
  Concentration of TS-142 and its metabolites in plasma
Step2; Subjective Alertness via Karolinska Sleepiness Scale (KSS) | Day 1 up to Day 8
  Step2; as a measure of subjective alertness which is scored by 10 cm-VAS scale ranging from 1, extremely alert, to 9, extremely sleepy at the next morning after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Sumida Hospital, Sumida-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kambe D, Hasegawa S, Imadera Y, Mano Y, Matsushita I, Konno Y, Ogo H, Uchimura N, Uchiyama M. Pharmacokinetics, pharmacodynamics and safety profile of the dual orexin receptor antagonist vornorexant/TS-142 in healthy Japanese participants following single/multiple dosing: Randomized, double-blind, placebo-controlled phase-1 studies. Basic Clin Pharmacol Toxicol. 2023 Nov;133(5):576-591. doi: 10.1111/bcpt.13930. Epub 2023 Sep 10. PMID 37563858